CLINICAL TRIAL: NCT02491853
Title: The Gulf Implantable Cardioverter-Defibrillator Registry (GulfICD)
Brief Title: The Gulf Implantable Cardioverter-Defibrillator Registry
Acronym: GulfICD
Status: Completed | Type: Observational
Sponsor: Gulf Heart Association (Other)
Collaborators: Medtronic (Industry); Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: GulfICD
Record Dates: First submitted 2015-07-01; First posted 2015-07-08 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Implantable Defibrillator User
MeSH Terms: interventions — Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Implantable Cardioverter Defibrillator — Implantable Cardioverter Defibrillator
  Other Names: ICD

SUMMARY:
This is a prospective observational multi-center multi-national study of the characteristics and outcomes of patients receiving implantable cardioverter-defibrillators (ICD) in the Arab Gulf region. A total of 1,500 patients will be enrolled. Data on baseline clinical characteristics, ICD programming parameters, inpatient outcomes, and clinical events such as mortality and ICD discharges over 1 year of follow-up will be collected.

DETAILED DESCRIPTION:
1. INTRUDUCTION 1.1 Background and Rationale The implantable cardioverter-defibrillator (ICD) is an effective tool for the prevention of sudden cardiac death (SCD) in high-risk patients. The efficacy of the ICD in the secondary and primary prevention of SCD was demonstrated in several large randomized clinical trials. The evolution of clinical trials of ICD therapy for primary prevention of SCD and the adoption of current national practice guidelines has lead to a considerable increase in the use of ICDs worldwide. In the Arab Gulf region, utilization of ICD therapy in high-risk patients had increased in the past decade with the arrival of trained electrophysiologists in the Gulf states. While observational studies in the United States and Europe have evaluated ICD use in those regions, there are scarce data on how ICDs are being used in the Gulf. Few single center studies have reported early results, and to date there are no prospective multinational data on ICD use in the Gulf. The Gulf Implantable Cardioverter-Defibrillator Registry (GulfICD) will be the first prospective, multicentre, multinational, observational studies of patients receiving ICDs in the Arab Gulf states.
2. STUDY OBJECTIVES AND ENDPOINTS The primary objective of the study is to describe the characteristics and outcomes of patients receiving ICD in the Arab Gulf region. Once completed, the data collected from GulfICD will be available for further secondary analyses including a description of ICD implant indications and programming patterns in the Gulf. As this is an observational and descriptive study, no specific endpoint is considered primary. However, main outcomes to be measured include all-cause mortality and ICD discharges including appropriate discharges for ventricular tachyarrhythmias and inappropriate discharges for other causes. Other endpoints to be measured include adverse events in the immediate post-implant period.
3. STUDY DESIGN Gulf ICD is a prospective, multicentre, multinational observational study.
4. SUBJECT SELECTION 4.1 Inclusion Criteria All adult patients 18 years or older, receiving a new ICD implant and willing to sign a consent form will be eligible.

   4.2 Exclusion Criteria Patients < 18 years and those not willing to sign a consent form. Subjects with existing ICDs undergoing pulse generator replacements or system revisions will not be included.
5. STUDY TREATMENTS All subjects will be treated per routine clinical practice. There will be no study-specific interventions/treatments.
6. STUDY PROCEDURES 6.1 Subject Withdrawal Subjects will have the right to withdraw from the study at anytime.
7. DATA VARIABLES 7.1 Data Variables Data variables to be collected are detailed in the attached case-report form(CRF) (Baseline CRF Appendix 1, Follow Up CRF Appendix 2). Data will be collected on paper CRF and then entered online. Variables to be collected at baseline will include the following domains: 1. Baseline Demographics, 2. Admission Characteristics, 3. Medical History and Risk Factors, 4. Diagnostic Procedures, 5. ICD Implant Procedure Characteristics, 6. ICD Programming, 7. Adverse Events, 8. Discharge Characteristics, 9. Discharge Medications, 10. Interim Events (during follow up).

   Variable definitions will be based on the American College of Cardiology/American Heart Association/Heart Rhythm Society 2006 Key Data Elements and Definitions for Electrophysiological Studies and Procedures and the American College of Cardiology National Cardiovascular Data Registry (NCDR) ICD Registry data dictionary (httpp://www.ncdr.com/Web NCDR/docs/public-data-collection-documents/icd_v2_datadictionary_codersdictionary_2-1.pdf?sfvrsn=2)
8. ADVERSE EVENT REPORTING 8.1 Adverse Events Reporting Since there will be no study-specific intervention/treatment, we do not expect study specific adverse events. However, adverse events that may be related to ICD implantation will be collected as per the attached CRF (Appendix 1).
9. DATA ANALYSIS 9.1 Sample Size Considerations Unlike randomized controlled trials where specific hypotheses are tested and primary comparative analyses are planned, observational studies and patient registries typically address descriptive objectives. Such objectives do not lend themselves to classic sample size/power calculations. Nonetheless, sample size considerations are important in the planning of registries. Typically, adequate sample size is required to ensure adequate precision around key outcomes and provide sufficient generalizability. With that in mind, we wanted to ensure adequate precision around two key outcomes: all-cause mortality and/or rate of appropriate ICD discharges at one year. To estimate an event rate of 10% at 1 year with a margin of error of 2% and 95% confidence intervals, a sample size of 829 patients is required. Since there is little guidance in the literature on such event rates among ICD recipients in the Gulf, and to compensate for losses to follow-up, we adjusted our sample size upwards to 1,000 patients. Sample size was later increased to 1,500 patients as additional funding became available. Such a sample size was considered logistically feasible given our experience with ICD implant rates in the Gulf.

   9.2 Statistical Methods Standard descriptive statistics will be used to analyse the data. Continuous variables will be summarized using mean and standard deviation or median and 25th and 75th percentile when significant deviation from a normal distribution is observed. Categorical variables will be summarized using counts and percentages. Basic univariate comparisons will be performed using Student's t-test or the Wilcoxon rank sum test as appropriate for continuous variables, and the Chi square test for categorical variables. Associations between baseline variables and outcomes during follow-up will be assessed using logistic regression or when exact event dates are available Cox proportional hazard models.
10. QUALITY CONTROL AND QUALITY ASSURANCE There is no substitute for good conscious. The investigators and their personnel filling the CRFs are responsible for filling the forms honestly and accurately. All forms must be filled prospectively. Quality control checking mechanisms are implemented in the online CRF system to prevent entry of inconsistent variables.
11. DATA HANDLING AND RECORD KEEPING 11.1 Case Report Forms/Electronic Data Records A CRF is required and should be collected and completed for each patient. Online data entry of the CRF will be available.

    11.2 Record Retention Investigators will retain the paper CRFs per local ethics regulations. Paper CRFs will be stored in a secure area with access only available to study investigators. The online CRF portal will be password protected.
12. ETHICS 12.1 Institutional Review Board/Ethics Committee Approval It is the responsibility of the investigator to get prospective approval of the study protocol, consent form, and any amendments from the local institutional review boards/ethic committee.

    12.2 Ethical Conduct of the Study The study will be conducted in accordance with the protocol and applicable local regulatory requirements and laws. Study conduct will also conform to the Declaration of Helsinki on Ethical Principles for Medical Research Involving Human Subjects adopted by the General Assembly of the World Medical Association

    12.3 Subject Information and Consent All investigators will ensure protections of subjects' personal data and subject names or identifiers will not be included on any reports or publications from the study. Each study subject will be informed about the study objectives and procedures and all questions will be answered. Subjects will have to sign a consent form to be enrolled in the study. The consent form must be in compliance with local regulatory requirements.
13. SPONSORSHIP GulfICD will be conducted under the auspices of the Gulf Heart Rhythm Society (GHRS) and the Gulf Heart Association (GHA). Partial funding for the development of the online CRF portal is provided by Medtronic, Inc.
14. STUDY STRUCTURE AND TIMELINE 14.1 Principal Investigators and Steering Committee Members The study co-principal investigators are: Dr Alawi Alsheikh-Ali, Dr Ahmad Hersi and Dr Adel Khalifa. Country-level Principal Investigators include: Dr Najib Alrawahi (Principal Investigator Gulf ICD-Oman), Dr Nidal Asaad (Principal Investigator Gulf ICD-Qatar), additional steering committee members at the time of this righting are: Dr Fayez Bokhari, Dr Ahmad Alfaqih and Dr Amin Daoulah (Kingdom of Saudi Arabia), Dr Fawzieh Alkandari (Kuwait), Dr Salim Al-Kaabi, Dr Omer Elhag, Dr Hani Sabbour and Dr Hosam Zaky (United Arab Emirates). Additional members will be added to the steering committee as more centers join the study.

    14.2 Study Timeline

    Below is a tentative study timeline:

    Milestone Date Initial talks between GHRS and Medtronic October 2011 Formal solicitation of funding submitted to Medtronic April 2012 Funding approved by Medtronic June 2012 Contract Signed with software company to develop online CRF system November 2012 Draft protocol and CRF circulated to Steering Committee December 2012 Development of online CRF portal and finalizing protocol December 2012-July 2013 Final protocol and CRF approved by steering committee August 2013 Submit for Institutional Review Board(IRB) approvals August/September 2013 Pilot online CRF September/October 2013 Official study launch November 2013 Submit "Methodology manuscript" December 2013 Complete enrolment November 2014 Complete follow-up for all patients November 2015 Data cleaning throughout study duration Data lockout January 2016 Start data analysis January 2016 Draft "main results manuscript" March 2016 Submit "main results manuscript" May 2016 Drafting and submissions of other manuscripts May 2016 onwards
15. PUBLICATION OF STUDY RESULTS Results of GulfICD will be disseminated through peer-reviewed manuscripts, abstracts, and presentations. The co-principal investigators and steering committee will be solely responsible for analysis, writing, and decision to submit for publications/presentation of all abstracts and manuscripts. Members of the steering committee will be co-authors on all study manuscripts that utilize the shared registry data. Manuscripts/abstracts based on country- or site-level data will require co-authorship by all steering committee members from the relevant country or site. Outside co-authors will be included if they meet the authorship requirements per the guidelines established by the International Committee of Medical Journal Editors and outlined in "Uniform Requirements for Manuscripts Submitted to Biomedical Journals; http://www.icmje.org/ethical_1author.html".

ELIGIBILITY:
Inclusion Criteria:

* New implantable cardioverter defibrillator
* Written consent

Exclusion Criteria:

* Pulse generator replacements or system revisions
* Failure to obtain written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient receiving de nove implantable cardioverter defibrillator for primary or secondary prevention of sudden cardiac death
Sampling Method: Non-Probability Sample
Enrollment: 1545 (Actual)
Dates: Start 2014-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
All-Cause Mortality | One Year

SECONDARY OUTCOMES:
Appropriate ICD Discharge | One Year
Inappropriate ICD Discharge | One Year
ICD Malfunction | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Alawi A. Alsheikh-Ali, MD, Principal Investigator — Sheikh Khalifa Medical City, Abu Dhabi, UAE; Ahmad S. Hersi, MD, Principal Investigator — King Saud University, Riyadh, KSA; Adel Khalifa, MD, Principal Investigator — Bahrain Defence Force Hospital, Manama, Bahrain
Locations (1):
- Sheikh Khalifa Medical City, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alsheikh-Ali AA, Hersi AS, Hamad AK, Al Fagih AR, Al-Samadi FM, Almusaad AM, Bokhari FA, Al-Kandari F, Al-Ghamdi BS, Al Rawahi N, Asaad N, Alkaabi S, Daoulah A, Zaky HA, Elhag O, Al Hebaishi YS, Sweidan R, Alanazi H, Chase D, Sabbour H, Al Meheiri M, Al Abri I, Amin M, Dagriri K, Ahmed AO, Shafquat A, Khan SH. The Gulf Implantable Cardioverter-defibrillator Registry: Rationale, Methodology, and Implementation. Heart Views. 2015 Oct-Dec;16(4):125-30. doi: 10.4103/1995-705X.172193. PMID 26900416